CLINICAL TRIAL: NCT07108166
Title: A Randomized, Single (Operator)-Blinded, Controlled Clinical Study for Assessing Major Symptoms and Function in Patients With Chronic Obstructive Pulmonary Disease (COPD) With Chronic Bronchitis Who Switch From Combustible Cigarettes (CIG) to Tobacco Heating System (THS)
Brief Title: Symptoms and Functions in Patients With COPD and Chronic Bronchitis Switching From CIG to THS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P1-FAF-16
Record Dates: First submitted 2025-05-22; First posted 2025-08-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: COPD; Smoking; Tobacco Use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cigarette (Active Comparator)
  Interventions: Other: Cigarette
- THS (Active Comparator)
  Interventions: Other: THS

INTERVENTIONS:
Other: Cigarette — COPD patients will continue to smoke their cigarettes ad libitum, with no brand restrictions.
  Arms: Cigarette
Other: THS — COPD patients will switch from cigarette smoking to ad libitum THS use, with no flavor variant restrictions.
  Arms: THS

SUMMARY:
The purpose of this randomized study is to demonstrate direct clinical benefit, i.e., observed benefits in how humans with COPD feel in terms of symptoms (e.g., cough frequency, shortness of breath, and other respiratory symptoms) and function (e.g., lung function, and six-minute walking test [6MWT]) after switching to THS compared to continuing to smoking cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Adult, both sexes, aged ≥ 40 years.
* Patient has read, understood, and signed the written informed consent form (ICF), which has received IEC or IRB approval.
* Patient with body mass index (BMI) 17.6-40.0 kg/m2 and body weight > 50 kg (male) or > 40 kg (female). Checked at V1 and V2.
* Patient has a CIG smoking history ≥ 10 years.
* Patient has been smoking ≥ 10 commercially available and/or roll-your-own CIG/day on average (no brand restriction) for at least the last year (based on self-reporting). Smoking status will be verified by Urine cotinine test (UCOT) ≥200 ng/mL. Intermittent CIG smoking abstinence, with or without Smoking Cessation Treatment during these attempts, not exceeding 10 days total within the past year will be allowed. Checked at V1 and V2.
* Patient has been advised to quit smoking, informed of smoking risks and of cessation programs as per SoC at V2, and is not willing to quit CIG use for the study duration. Checked at V1 and V2.
* Patient agrees to be randomized into one of the two study arms. Checked at V2.
* Patient with confirmed COPD via spirometry performed at V1 (FEV1/FVC <70%, post-bronchodilator (-BD)) and COPD severity classified by the Global Initiative for Chronic Obstructive Lung Diseases (GOLD) as GOLD 2 or 3 (30%≤ FEV1 < 80% predicted, -BD) with presence of chronic bronchitis (cough and mucus most of the days for > three months a year for the two consecutive years prior to the screening visit). Checked at V2.
* Patient has cough frequency of ≥ 10 cough/hour during daytime from objective count sensor applied at V1, used to verify eligibility at V2. (Daytime is defined as occurring between 07:00:00 and 22:59:59, based on the local time zone of the site where the patient is assessed.)

Exclusion Criteria:

* Patient who self-report concomitant daily use of inhaled cannabis or any type of nicotine containing products other than CIG within the last year.
* Patient with COPD (moderate or severe) exacerbation that has not resolved according to the GOLD standard (e.g., requirement of additional therapy) or investigator's discretion. Checked at V1 and V2.
* Patient with currently active cancer or history of any cancer within the last 5 years prior to V1, except for those with basal cell carcinoma of the skin.
* Patient with acute worsening symptoms of chronic bronchitis or other active respiratory or systemic infections that have not resolved. Checked at V1 and V2.
* Patient with medical condition(s) that would jeopardize his(her) safety in the context of this study (e.g., safety laboratory parameters, abnormal ECG) or with a condition that would jeopardize study results (e.g., gastroesophageal reflux disease (GERD), heart failure, severe chronic lung emphysema, active symptomatic hay fever), as per Investigator's discretion. Checked at V1 and V2.
* Patient is legally incompetent, physically, and/or mentally incapable of giving consent (e.g., emergency situation, under guardianship, in a social or sanitary establishment, prisoner or involuntarily incarcerated, unable to read).
* Patient with a history of asthma.
* Employee of the investigational site or any other party involved in the study, or their first-degree relatives (parent, child, spouse).
* Current or former employee of the tobacco or e-cigarette industry or their 1st-degree relatives.
* Patient with active or history of alcohol and/or drug abuse within the past year.
* Patient with positive serological tests for human immunodeficiency virus (HIV) 1/2, hepatitis B or C (Hep B/C).
* Patient with any concomitant issues (e.g., medical, psychiatric, and/or social reason) that, as per Investigator's discretion, would place the study patient at an unacceptable risk for participation in the study.
* Patient who participated in any trial (for investigational medicine, or other type of intervention) that may have interfered with COPD disease progression and symptoms (including cough and dyspnea) within the last three months as per investigator's discretion.
* Patient using any systemic (injectable or oral) corticosteroids (acute or chronic treatments) or oxygen therapy in the last 2 months excluding short term use for a COPD exacerbation.
* Patient currently being treated with angiotensin-converting enzyme (ACE) inhibitors or opioids, or those who have used ACE inhibitors within 4 weeks or opioids within 1 week prior to screening. Checked at V1 and V2.
* Patient treated with biologic therapies for COPD (e.g., Dupilumab) in the last 6 months.
* Female patient is pregnant, breastfeeding or lactating, or anticipating becoming pregnant withing the duration of the study. Checked at V1 and V2.
* Female of childbearing potential who is capable of getting pregnant, defined as a female patient who does not agree to use an acceptable method of effective contraception during the entire study, a female patient that is not surgically sterilized (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year). Checked at V1 and V2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in 24-hour cough frequency | Measured from start of product use to end of week 24 (end of the exposure period).
  To demonstrate a change in 24-hour cough frequency in COPD patients with chronic bronchitis switching from cigarette (CIG) to THS compared to those who continue to smoke CIG.

SECONDARY OUTCOMES:
Changes in lung function (from Baseline in FEV1 post-bronchodilator) | Measured from start of product use to end of week 24 (end of the exposure period).
  To describe changes from Baseline in FEV1 post-bronchodilator in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Changes in the 24-hour cough frequency over time | Measured from start of product use to 12 weeks, at the end of weeks 1, 4, and 12.
  To describe changes in the 24-hour cough frequency over time in in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Percentage of patients with a change in 24-hour cough frequency over time | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24
  To describe the percentage of patients with a change in 24-hour cough frequency over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Changes in the Cough Quality of Life Questionnaire (CQLQ) on chronic cough | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  To describe changes in the Cough Quality of Life Questionnaire (CQLQ) on chronic cough in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG. It consists of 28 items to which the patient responds on a 4-point Likert scale, ranging from 1=strongly disagree, to 4=strongly agree. The total score is the sum of all individual items. Lower scores indicate a better outcome.
Changes in cough severity over time | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  To describe changes in cough severity over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Changes in bronchial hyperresponsiveness (BHR) mannitol test over time | Measured from start of product use to end of week 24 (end of the exposure period).
  To describe changes in bronchial hyperresponsiveness (BHR) mannitol test over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG, at sites with full testing capabilities for BHR testing.
Impact of COPD (cough, sputum, dyspnea, chest tightness) on health status | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  To assess the impact of COPD (cough, sputum, dyspnea, chest tightness) on health status in COPD by the COPD Assessment Test (CAT) over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
  The CAT questionnaire consists of eight items, each answered on a semantic six-point differential scale from 0 to 5. The CAT score is calculated as the sum of the responses. Scores range from 0 to 40 with higher scores representing worse health outcomes.
Changes in shortness of breath assessed over time | Measured from start of product use to end of week 24 (end of the exposure period).
  To describe changes in shortness of breath assessed over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Changes in functional capacity over time | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 12 and 24.
  To describe changes in functional capacity over time in COPD patients with chronic bronchitis switching from CIG to THS compared to those who continue to smoke CIG.
Changes in exposure to carbon monoxide over time | Measured from start of product use to end of week 24 (end of the exposure period).
  Change from Baseline in carbon monoxide (CO) exposure levels measured from venous blood carboxyhemoglobin (COHb) at the end of weeks 1, 4, 12, and 24.
Changes in self-reported tobacco and nicotine containing product consumption | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  Changes from Baseline in self-reported tobacco and nicotine containing product consumption and change in self-reported CIG and overall tobacco consumption evaluated with the ABOUT Tobacco exposure Tool (ABOUT-TeT). This instrument is a questionnaire to record self-reported consumption of tobacco and nicotine containing products. Patients will be asked to self-report the number of CIG, THS Induction Sticks, and other tobacco and nicotine containing products used on average per day over the last week. Patients will complete the questionnaire every seven days, from week 1 to week 24.
Changes in nicotine exposure levels | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  Change from Baseline in nicotine exposure levels in spot urine adjusted to creatinine (Nicotine equivalents [NEQ]).
Changes in acrylonitrile exposure levels | Measured from start of product use to 24 weeks (end of the exposure period), at the end of weeks 1, 4, 12, and 24.
  Change from Baseline in acrylonitrile exposure levels in 2-Cyanoethyl Mercapturic Acid N-Acetyl-S-(2-cyanoethyl)-L-cysteine (2-CyEMA) measured in urine and expressed as concentration adjusted to creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jaumont, MD, Study Chair — Philip Morris Products S.A.
Locations (111):
- United States (44):
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Florida International Medical Research, Coral Gables, Florida
  - Alfa Medical Research, Davie, Florida
  - Omega Research Debary, LLC, DeBary, Florida
  - D&H Doral Research Center, Doral, Florida
  - Felicidad Med Research, Hialeah, Florida
  - The Medici Medical Research, LLC, Hollywood, Florida
  - D&H Pompano Research Center, Margate, Florida
  - Med-Care Research Corp, Miami, Florida
  - EMDA Clincal Research, Miami, Florida
  - Sones Medical Research, Miami, Florida
  - Suncoast Research Group, LLC dba Flourish Research, Miami, Florida
  - Melgar-Caro Medcenter and Community Research, Miami, Florida
  - D&H National Research Center- Miami, Miami, Florida
  - Biomed Research & Medical Center.Llc, Miami, Florida
  - Global Health Clinical Trials Corp., Miami, Florida
  - Professional Research Center Inc, Miami, Florida
  - Newgen Health Group, Miami, Florida
  - Reserka LLC, Miami, Florida
  - Pharma Medical Innovations, Miami Lakes, Florida
  - San Marcus Research, Miami Lakes, Florida
  - MedQuest Translational Sciences LLC, Miami Lakes, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Comprehensive Medical & Research Center, Plantation, Florida
  - CDC Research Institute, Port Saint Lucie, Florida
  - Treasure Coast Medical Research Group, Port Saint Lucie, Florida
  - Advanced Research Institute, Inc, St. Petersburg, Florida
  - D&H Tamarac Research Center, Tamarac, Florida
  - Metropolitan Clinical Research Center, Tamarac, Florida
  - Optimum Clinical Trial Group, Tampa, Florida
  - Pivotal Research Solutions, Stonecrest, Georgia
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - HDH Research Inc, Houston, Texas
  - Prolato Research LLC., Houston, Texas
  - Houston Pulmonary Medicine Associates, Houston, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
  - Accurate Clinical Research, Inc., Humble, Texas
  - Metroplex Pulmonary & Sleep Center, McKinney, Texas
  - Element Research Group, San Antonio, Texas
  - Medrasa Clinical Research, Sherman, Texas
  - Pulmonics Plus, Waxahachie, Texas
- Bulgaria (6):
  - MHAT Rahila Angelova, Pernik
  - MHAT Lyulin EAD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Pulmovision Ltd, Sofia
  - SHATPD Dr. Treyman, Veliko Tarnovo
  - SHATPPD Vratsa, Vratsa
- Czechia (6):
  - MUDr. Otakar Hokynar - plicni ambulance, Kralupy nad Vltavou
  - Ordinace pro tbc a respirační nemoci s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - Medicon a.s., Prague
  - Prvni plicni ambulance s.r.o., Prague
  - Pneumologie Varnsdorf s.r.o., Varnsdorf
- Germany (14):
  - Klinische Forschung Berlin Mitte /Pratia Germany, Berlin
  - Research Center for Medical Studies, Berlin
  - Klifeck GmbH, Delitzsch
  - Klinische Forschung Hannover-Mitte GmbH /Pratia Germany, Hanover
  - Klinische Forschung Karlsruhe GmbH / Pratio Germany, Karlsruhe
  - Facharzt für Innere Medizin und Pneumologie, Leipzig
  - POIS Sachsen GmbH, Leipzig
  - Ballenberger Freytag Wenisch - Institut für klinische Forschung GmbH, Neu-Isenburg
  - FutureMeds Frankfurt, Offenbach
  - Praxis Reinfeld Mitte, Reinfeld
  - Siteworks - Prüfzentrum Schleswig | RespiRatio, Schleswig
  - BAG Peter Fried / Dr. med. Roman Rubin, Wiesbaden
  - Velocity Clinical Research Wiesbaden, Wiesbaden
  - Lungenpraxis Witten, Witten
- Japan (9):
  - Soejima Clinic, Fukuoka
  - JCHO Nihonmatsu Hospital, Fukushima
  - Maebashi North Hospital, Gunma
  - Akashi Medical Center, Hyōgo
  - Fukuwa Clinic, Tokyo
  - Kouwa Clinic, Tokyo
  - Sanyuudo Hospital, Yamagata
  - Yokohama Minoru Clinic, Yokohama
  - Clinical Research Hospital Tokyo, Yotsuya
- Poland (10):
  - Centrum Medycyny Oddechowej Mroz Spolka jawna, Bialystok
  - BioResearch Group Sp. z.o.o, Kajetany
  - FutureMeds Krakowskie Centrum Medyczne, Krakow
  - FutureMeds Łódź, Lodz
  - AmiCare Centrum Medyczne, Lodz
  - RCMed Oddział Sochaczew, Sochaczew
  - FutureMeds Warszawa Centrum, Warsaw
  - FutureMeds Targówek, Warsaw
  - Dobrostan, Wroclaw
  - FutureMeds Wrocław, Wroclaw
- Romania (7):
  - Ames Research Center, Bragadiru
  - Sc. Centrul Medical Sana Srl, Brasov
  - Sana Medical Center, Bucharest
  - Ames Research Center, Călăraşi
  - Clintrial Medical Centre SRL, Dobrosloveni
  - Spital de Pneumologie dr Lavinia Davidescu Oradea, Oradea
  - AI Clinical Research, Sibiu
- Slovakia (5):
  - PANACEUM s.r.o., Košice
  - Vseobecna ambulancia pre dospelych, Košice
  - Pulmo s.r.o.,, Prešov
  - Plucna ambulancia Hrebenar S.R.O., Spišská Nová Ves
  - Alergia s. r. o., Topoľčany
- United Kingdom (10):
  - Panthera Biopartners, Enfield
  - Panthera Biopartners, Glasgow
  - Velocity High Wycombe, High Wycombe
  - 4 Medical Clinical Solutions (4MCS), London
  - 4 Medical Clinical Solutions (4MCS), Manchester
  - FutureMeds Liverpool, Metropolitan Borough of Wirral
  - Panthera Biopartners, Preston
  - Panthera Biopartners, Rochdale
  - Panthera Biopartners, Sheffield
  - Panthera Biopartners, York